CLINICAL TRIAL: NCT05643118
Title: Evaluation of the Safety and Tolerability of OLX10212 in Patients With Neovascular Age-Related Macular Degeneration
Brief Title: Evaluation of OLX10212 in Patients With Neovascular Age-related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Olix Pharmaceuticals, Inc. (Industry)
Collaborators: Trial Runners, LLC (Other); Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OLX10212-01
Record Dates: First submitted 2022-11-10; First posted 2022-12-08 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Neovascular age-related macular degeneration; OLX10212; siRNA; intravitreal injection; safety and tolerability; preliminary efficacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A 100 μg/eye/50 μL (Experimental): study eye treated with 100 μg (94.3 μg free acid) of OLX10212
  Interventions: Genetic: OLX10212 is a cell penetrating asymmetric small interference RNA (cp-asiRNA)
- Part A 250 μg/eye/50 μL (Experimental): study eye treated with 250 μg (235.8 μg free acid) of OLX10212
  Interventions: Genetic: OLX10212 is a cell penetrating asymmetric small interference RNA (cp-asiRNA)
- Part A 500 μg/eye/50 μL (Experimental): study eye treated with 500 μg (471.5 μg free acid) of OLX10212
  Interventions: Genetic: OLX10212 is a cell penetrating asymmetric small interference RNA (cp-asiRNA)
- Part A 750 μg/eye/50 μL (Experimental): study eye treated with 750 μg (707.3 μg free acid) of OLX10212
  Interventions: Genetic: OLX10212 is a cell penetrating asymmetric small interference RNA (cp-asiRNA)
- Part A 950 μg/eye/50 μL (Experimental): study eye treated with 950 μg (895.9 μg free acid) of OLX10212
  Interventions: Genetic: OLX10212 is a cell penetrating asymmetric small interference RNA (cp-asiRNA)
- Part B 750 μg/eye/50 μL (Experimental): study eye treated with a total of 3 intravitreal injections of 750 μg (707.3 μg free acid) of OLX10212 each 28 days apart
  Interventions: Genetic: OLX10212 is a cell penetrating asymmetric small interference RNA (cp-asiRNA)
- Part B 950 μg/eye/50 μL (Experimental): study eye treated with a total of 3 intravitreal injections of 950 μg (895.9 μg free acid) of OLX10212 each 28 days apart
  Interventions: Genetic: OLX10212 is a cell penetrating asymmetric small interference RNA (cp-asiRNA)

INTERVENTIONS:
Genetic: OLX10212 is a cell penetrating asymmetric small interference RNA (cp-asiRNA) — Clear colorless solution dissolved in 1X PBS and injected intravitreally
  Other Names: OLX10212

SUMMARY:
This is a Phase 1, multicenter, open-label, single- and multi-dose, dose-escalating study of OLX10212 in patients with neovascular age-related macular degeneration (AMD). This study is composed of 2 parts: Part A and Part B. Part A is a single ascending dose study, and Part B is a multiple ascending dose study. The primary objective is to evaluate the safety and tolerability of single and multiple intravitreal injection(s) of OLX10212 in patients with neovascular AMD. The exploratory objectives are to evaluate the preliminary efficacy of single and multiple intravitreal injection(s) of OLX10212 in patients with neovascular AMD, and to evaluate the pharmacokinetics (PK) of single and multiple intravitreal injection(s) of OLX10212 in patients with neovascular AMD.

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, open-label, single- and multi-dose, dose escalation study to evaluate the safety, tolerability, and preliminary efficacy of OLX10212 in the treatment of age-related macular degeneration (AMD). This study is composed of 2 parts: Part A and Part B. Part A is a single ascending dose study, i.e. participants will receive one intravitreal injection of OLX10212 at different dose levels and Part B is a multiple ascending dose study, i.e. participants will receive up to three intravitreal injections of OLX10212. Up to 42 individuals with AMD will be invited to participate in this study. The mechanism of action of OLX10212 holds promise to treat AMD by improving inflammation in the retina which is typically observed in patients with AMD. This is the first time OLX10212 is used in patients with AMD. Safety and tolerability of OLX10212 will be assessed via detailed ophthalmologic evaluations, vital signs, and clinical laboratory testing. In addition, plasma concentrations of OLX10212 will be measured and evaluations of the therapeutic effects of OLX10212 will be performed.

Part A uses a dose-ascending, sequential design to evaluate up to five doses of OLX10212, starting with the lowest dose of OLX10212 in a 50-μL injection. Up to six patients will be enrolled at each dose level. Each of the enrolled patients will receive a single intravitreal administration of OLX10212. The safety and tolerability evaluation period will encompass the first 14 days following OLX10212 administration. The effects of OLX10212 will be observed up to 24-weeks after injection. Based on the safety and tolerability evaluation, a decision will be made whether or not to increase the dose to the next higher dose levels for the subsequent patient cohorts. Therefore, a total of up to 30 patients (up to 5 dose levels and up to 6 patients/dose level) will be enrolled in Part A of this study.

Part B of this study uses a dose-ascending, sequential design to evaluate 2 dose levels of OLX10212 (750 and 950 μg/eye/50 μL), starting with the 750 μg/eye/50 μL dose. Three patients will initially be enrolled in each cohort. Each of the enrolled patients will receive a total of up to three intravitreal injections of OLX10212, each four weeks apart (Week 0, Week 4, and Week 8). The DLT evaluation period will encompass the first 10 weeks following the first OLX10212 administration (ending 2 weeks following the third OLX10212 administration), during which safety and tolerability will be assessed at each visit. In addition, the plasma concentrations of OLX10212 will be measured and therapeutic effects will be evaluated. A total of up to 12 patients with AMD (3 dose levels and up to 6 patients/dose level) will be invited to participate in Part B of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥50 years of age
2. Primary subfoveal CNV lesions secondary to AMD, including juxtafoveal lesions that affect the fovea, as evidenced by FA in the study eye
3. CNV must be ≥50% of the total lesion size in the study eye
4. ETDRS BCVA score ranging from 20/60 to 20/400 in the study eye
5. Clear ocular media and adequate pupillary dilation (able to dilate pupil to ≥4 mm using standard mydriatics) in the study eye to permit good stereoscopic fundus photography
6. Retinal thickness ≥200 μm in the macular region of the study eye as measured by SD-OCT, and active neovascular AMD, in the opinion of the Investigator
7. Willing, committed, and able to return for all clinic visits and complete all study-related procedures
8. Able to read (or if unable to read due to visual impairment, be read to verbatim by the person administering the informed consent or by a family member), understand, and willing to sign the informed consent form

Exclusion Criteria:

1. Any prior systemic treatment for neovascular AMD in either eye, except dietary supplements or vitamins or systemic anti-VEGF therapy, or planned use at any time during the study
2. Any prior treatment in the study eye with another investigational agent to treat neovascular AMD within 6 months prior to Day 0 or planned use at any time during the study
3. Prior treatment with anti-VEGF agents as follows:

   1. Anti-VEGF therapy in the study eye within 4 weeks prior to Day 0
   2. Anti-VEGF therapy in the study eye at any time to which there was no response, as defined by the presence of at least 1 of the following conditions: (1) persistent (plasma) fluid exudation, (2) unresolved or new hemorrhage, and (3) progressive lesion fibrosis
   3. Anti-VEGF therapy in the fellow eye with an investigational agent (not FDA approved, unless it is bevacizumab) within 3 months prior to Day 0 (prior treatment with an FDA approved anti-VEGF therapy in the fellow eye is allowed at any time)
   4. Systemic anti-VEGF therapy, investigational or FDA approved, within 3 months prior to Day 0 or planned use at any time during the study
4. Scar or fibrosis in the study eye involving >50% of the total lesion size
5. Retinal pigment epithelial tears or rips in the study eye involving the macula within 6 months prior to Day 0
6. History of any vitreous hemorrhage in the study eye within 4 weeks prior to Day 0
7. Presence of other causes of CNV in the study eye, including pathologic myopia, ocular histoplasmosis syndrome, angioid streaks, choroidal rupture, or multifocal choroiditis
8. Clinical evidence of moderate or severe diabetic retinopathy, diabetic macular edema, or any other inflammatory or occlusive vascular disease affecting the retina (other than AMD) in either eye
9. History of stage ≥2 macular hole in the study eye
10. Any prior intraocular or periocular surgery on the study eye within 3 months prior to Day 0 (lid surgery is allowed if it took place at least 1 month prior to Day 0 and is unlikely to interfere with OLX10212 injection). Prior vitrectomy in the study eye, surgery for retinal detachment in the study eye, and prior trabeculectomy or other filtration surgery in the study eye are not permitted at any time
11. Uncontrolled glaucoma (defined as IOP ≥25 mmHg despite treatment with antiglaucoma medication) in the study eye
12. Glaucoma in the study eye requiring treatment with 3 or more antiglaucoma medications
13. Active intraocular inflammation or history of uveitis in either eye
14. Presence or history of ocular or periocular infection in either eye within 2 weeks prior to Day 0
15. Presence of scleromalacia in the study eye
16. Aphakia or absence of posterior capsule in the study eye (unless due to yttrium aluminum garnet [YAG] posterior capsulotomy)
17. Prior therapeutic radiation in the region of the study eye or planned use at any time during the study
18. Significant media opacities, including cataract, in the study eye that, in the opinion of the Investigator, could interfere with visual acuity, assessment of safety, or fundus photography
19. Any concurrent intraocular condition in the study eye (eg, cataract) that, in the opinion of the Investigator, could (1) require either medical or surgical intervention during the 24- or 32-week study period (Part A or Part B, respectively), (2) increase the risk to the patient beyond what is to be expected from standard intraocular injection procedures, or (3) otherwise interfere with the injection procedure or efficacy or safety evaluation
20. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that might affect interpretation of the results of the study or renders the patient at high risk for treatment complications
21. Participation as a patient in any clinical study or prior systemic or ocular treatment with an investigational agent within 12 weeks prior to Day 0
22. Prior systemic or intraocular treatment with long-acting steroids within 6 months prior to Day 0 or planned use at any time during the study
23. History of allergy to povidone iodine
24. Known allergy to fluorescein sodium for injection in angiography
25. Unwillingness among females who are pregnant, breastfeeding, or of childbearing potential to practice adequate contraception throughout the study. Adequate contraceptive measures include oral contraceptives (stable use for ≥2 cycles prior to Day 0), intrauterine device, Depo-Provera® (Pfizer, Inc., New York) or Norplant System® (Pfizer, Inc., New York) implants, bilateral tubal ligation, vasectomy, and condom or diaphragm plus contraceptive sponge, foam, or jelly. A female is considered to be of childbearing potential unless she is premenstrual, 1 year postmenopausal, or 3 months post-surgical sterilization. All females of childbearing potential, including those with post-tubal ligation, must have a negative urine pregnancy test result at Day 0 and every 4 weeks as outlined in the Schedule of Activities. A negative serum pregnancy test must be obtained at Screening.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Best-corrected visual acuity (BCVA) | 28 days after last dose administration
  Visual acuity using an ETDRS chart
Intraocular pressure (IOP) | 28 days after last dose administration
  Millimeters of mercury (mmHg)
Slit lamp | 28 days after last dose administration
  Anterior segment of the eye examination
Fundus examination | 28 days after last dose administration
  Posterior segment of the eye examination
Spectral-domain optical coherence tomography (SD-OCT) | 28 days after last dose administration
  Evaluation of retinal characteristics
Fluorescein angiography (FA) | 28 days after last dose administration
  Evaluation of retinal vasculature

OTHER OUTCOMES:
Spectral-domain optical coherence tomography | Week 24
  Changes in retinal thickness and relative changes (%) in CNV lesion area (mm2)
Fluorescein angiography | Week 24
  Changes in retinal fluid and relative changes (%) in CNV lesion area (mm2)
Cmax | Day 0, Day 1, Day 2, and Day 3 for Part A and Day 0, Day 1, Day 2, Day 3, Day 28, Day 29, Day 30, Day 31,Day 56, Day 57, Day 58, and Day 59 for Part B
  Peak plasma concentration of OLX10212
Tmax | Day 0, Day 1, Day 2, and Day 3 for Part A and Day 0, Day 1, Day 2, Day 3, Day 28, Day 29, Day 30, Day 31,Day 56, Day 57, Day 58, and Day 59 for Part B
  Time at which Cmax occurs
AUC | Day 0, Day 1, Day 2, and Day 3 for Part A and Day 0, Day 1, Day 2, Day 3, Day 28, Day 29, Day 30, Day 31,Day 56, Day 57, Day 58, and Day 59 for Part B
  Total area of plasma concentration of OLX10212

CONTACTS AND LOCATIONS:
Overall Officials: Toni Bransford, MD, Study Director — Olix Pharmaceuticals, Inc.
Locations (5):
- United States (5):
  - California Retina Consultants, Santa Maria, California
  - University Retina, Oak Forest, Illinois
  - The Retina Institute, St Louis, Missouri
  - Ophthalmic Consultants of the Capital Region, Troy, New York
  - Texas Retina Consultants, Bellaire, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hwang J, Chang C, Kim JH, Oh CT, Lee HN, Lee C, Oh D, Lee C, Kim B, Hong SW, Lee DK. Development of Cell-Penetrating Asymmetric Interfering RNA Targeting Connective Tissue Growth Factor. J Invest Dermatol. 2016 Nov;136(11):2305-2313. doi: 10.1016/j.jid.2016.06.626. Epub 2016 Jul 15. PMID 27427487